CLINICAL TRIAL: NCT01226316
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD5363 Under Adaptable Dosing Schedules in Patients With Advanced Solid Malignancies
Brief Title: Safety, Tolerability & Potential Anti-cancer Activity of Increasing Doses of AZD5363 in Different Treatment Schedules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3610C00001; EudraCT number: 2010-022167-35; 2010-022167-35 (EudraCT Number)
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Malignancy; Safety and Tolerability; Pharmacokinetics; Pharmacodynamics; Tumour Response; Advanced or Metastatic Breast Cancer; Ovarian Cancer; Cervical Cancer; Endometrial Cancer; PIK3CA; AKT1; PTEN; ER Positive; HER2 Positive
Keywords: Advanced solid malignancy,PIK3CA mutated,AKT1 mutated, PTEN mutation, PTEN alteration, metastatic,ER+,breast,ovarian,endometrial,AZD5363,AKT inhibitor,
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A and B Schedule 1, Continuous dosing (Experimental): Part A: Ascending doses of AZD5363 administered orally, every day to define the maximum tolerated dose. Part B: Dose expansion phase, at the defined maximum tolerated dose or recommended dose from Part A.
  Interventions: Drug: AZD5363
- Parts A,B,C,D Schedule 2, Intermittent dosing (Experimental): Part A: Ascending doses of AZD5363 administered orally, twice daily, on a 7-day repeating regimen (4 days on, 3 days off and 2 days on, 5 days off), to define the maximum tolerated dose. Part B: Dose expansion phase, at the defined maximum tolerated dose or recommended dose from Part A (4 days on, 3 days off and 2 days on, 5 days off). Part C and D: AZD5363 orally, twice daily on an intermittent regimen (4 days on, 3 days off).
  Interventions: Drug: AZD5363
- Parts A and B Schedule 3, Intermittent dosing. (Experimental): Part A: Ascending doses of AZD5363 administered orally, twice daily, on an alternative weekly regimen. Initiation of Schedule 3 is dependant on emerging clinical data.
  Part B: Dose expansion phase, at the defined maximum tolerated dose or recommended dose from Part A
  Interventions: Drug: AZD5363
- Parts E and F, Intermittent dosing with Fulvestrant (Experimental): Oral AZD5363 twice daily, 4 days on treatment, 3 days off treatment to cessation of therapy combined with background therapy of fulvestrant at its licensed dose of 500mg intramuscularly on days 1,15,29 and once monthly thereafter to cessation of therapy.
  Interventions: Drug: AZD5363

INTERVENTIONS:
Drug: AZD5363 — Patients will receive a single dose of AZD5363, administered orally, followed by a 3-7 day wash-out period. Patients will then commence with twice-daily dosing, administered orally, every day, to cessation of therapy.
  Arms: Part A and B Schedule 1, Continuous dosing
Drug: AZD5363 — Patients will be given AZD5363 administered orally as a single dose, followed by a 3-7 day wash-out period. Patients will then receive AZD5363 twice daily on 6 or fewer days per weekly regimen, to cessation of therapy. Parts C,D: Oral AZD5363 twice daily, 4 days on treatment, 3 days off treatment, to cessation of therapy.
  Arms: Parts A,B,C,D Schedule 2, Intermittent dosing
Drug: AZD5363 — Optional additional schedule. Patients will be given AZD5363 administered orally. Regimen to be determined in response to emerging clinical findings.
  Arms: Parts A and B Schedule 3, Intermittent dosing.
Drug: AZD5363 — Patients will receive oral AZD5363 twice daily (4 days on 3 days off treatment)combined with background therapy of fulvestrant at licensed dose of 500mg intramuscularly on days 1,15,29 and once monthly thereafter.
  Arms: Parts E and F, Intermittent dosing with Fulvestrant

SUMMARY:
This study is designed to investigate the safety and tolerability of a new drug, AZD5363, in patients with advanced cancer - and to identify a dose and schedule that can be used in the future. This study will also investigate how the body handles AZD5363 (ie, how quickly the body absorbs and removes the drug). This study will also investigate anti-tumour activity of AZD5363 in patients with advanced / metastatic breast, gynaecological cancers or other solid cancers bearing either AKT1 / PIK3CA or PTEN mutation.

DETAILED DESCRIPTION:
A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD5363 under Adaptable Dosing Schedules in Patients with Advanced Solid Malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* Parts A,B: The presence of a solid, malignant tumour, excluding lymphoma, that is resistance to standard therapies or for which no standard therapies exist.
* ER+/HER2+ breast, ovarian, cervical, endometrial cancer, or other solid cancers, resistance to standard therapies with a PIK3CA gene mutation (Part C), AKT1 gene mutation (Part D) or a dysregulatory aberration on the PIK/AKT pathway (Part D), advanced or metastatic ER+ positive breast cancer that has an AKT1 gene mutation (Part E) or advanced or metastatic ER+ positive breast cancer that has a PTEN gene mutation (Part F).
* The presence of at least one lesion that can be accurately assessed at baseline by CT, MRI or plain X-ray and is suitable for repeated assessment. Estimated life expectancy of more than 12 weeks.
* Estimated life expectancy of more than 12 weeks.

Exclusion Criteria:

* Clinically significant abnormalities of glucose metabolism.
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable (not requiring steroids).
* Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and HIV.
* Evidence of clinically significant cardiac abnormalities, uncontrolled hypotension, left ventricular ejection fraction below the lower limit of normal for the site or experience of significant cardiac interventional procedures.
* A bad reaction to AZD5363 or any drugs similar to it in structure or class.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Parts A,B,C,D,E & F : Safety and tolerability of AZD5363 in terms of adverse events and serious adverse events | Adverse events, serious adverse events and deaths will be collected from screening to 28 days after study drug discontinuation.
Parts A,B,C,D,E & F : Safety and tolerability of AZD5363 in terms of death | Deaths will be collected from screening to 28 days after study drug discontinuation
Parts A,B,C,D,E & F: Safety and tolerability of AZD5363 by assessing changes from baseline of laboratory data (clinical chemistry, haematology, urinalysis) | Laboratory data will be collected from screening to 28 days after study drug discontinuation
Parts A,B,C,D,E & F: Safety and tolerability of AZD5363 in terms of changes from baseline in vital signs and in electrocardiogram (ECG) parameters | Vital signs and ECGs will be recorded from screening to 28 days after study drug discontinuation
Parts A,B,C,D,E & F: Safety and tolerability of AZD5363 by assessing changes from baseline in electrocardiogram (ECG) parameters | ECGs will be collected from screening to 28 days after study drug discontinuation.
Parts A,B,C,D,E & F: Safety and tolerability of AZD5363 by assessing changes from baseline of glucose laboratory parameters (Urine, serum and plasma glucose, glycosylated haemoglobin). | Glucose parameters will be collected from screening to 28 days after study discontinuation.
Parts A,B,C,D,E & F: Safety and tolerability of AZD5363 by assessing left ventricular ejection fraction (LVEF). | Multiple Gated Acquisition (MUGA) or Echocardiogram assessments to be carried out from screening until study drug discontinuation

SECONDARY OUTCOMES:
To characterise AZD5363 PK following single & multiple dosing by assessment of maximum plasma concentration,time to Cmax, terminal rate constant, terminal half life,area under the plasma concentration-time curve,plasma clearance & volume of distribution. | Sample:Part A&B:Cycle0Day1(predose,30min,1,2,4,6,8,10-12,24&48h postdose),C1D1(predose),D8/Last wkly dose(predose,30min,1,2,4,6,8,10-12h postdose),D15/Last wkly dose+7(predose),Part C,D,E&F:C1D1(predose,2,4h postdose)&D11(predose,2,4h postdose)
Parts A,B,C,D,E&F: To obtain a preliminary assessment of anti-tumour activity of AZD5363 via use of Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 | Tumour assessment by RECIST at 6,12,18,24wks then at 12 weekly intervals until discontinuation of study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gaia Schiavon, MSD, Study Director — AstraZeneca; Udai Banerji, MD, PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (32):
- United States (11):
  - Research Site, Los Angeles, California
  - Research Site, Stanford, California
  - Research Site, West Hollywood, California
  - Research Site, Aurora, Colorado
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, København Ø, Denmark
- France (3):
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Villejuif
- Italy (3):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Prato
- Japan (4):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Sapporo
- Research Site, Amsterdam, Netherlands
- Research Site, Singapore, Singapore
- Spain (2):
  - Research Site, Madrid
  - Research Site, Valencia
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Smyth LM, Reichel JB, Tang J, Patel JAA, Meng F, Selcuklu DS, Houck-Loomis B, You D, Samoila A, Schiavon G, Li BT, Razavi P, Piscuoglio S, Reis-Filho JS, Taylor BS, Baselga J, Solit DB, Hyman DM, Berger MF, Chandarlapaty S. Utility of Serial cfDNA NGS for Prospective Genomic Analysis of Patients on a Phase I Basket Study. JCO Precis Oncol. 2021 Jan 8;5:PO.20.00184. doi: 10.1200/PO.20.00184. eCollection 2021. PMID 34250397
- [Derived] Smyth LM, Batist G, Meric-Bernstam F, Kabos P, Spanggaard I, Lluch A, Jhaveri K, Varga A, Wong A, Schram AM, Ambrose H, Carr TH, de Bruin EC, Salinas-Souza C, Foxley A, Hauser J, Lindemann JPO, Maudsley R, McEwen R, Moschetta M, Nikolaou M, Schiavon G, Razavi P, Banerji U, Baselga J, Hyman DM, Chandarlapaty S. Selective AKT kinase inhibitor capivasertib in combination with fulvestrant in PTEN-mutant ER-positive metastatic breast cancer. NPJ Breast Cancer. 2021 Apr 16;7(1):44. doi: 10.1038/s41523-021-00251-7. PMID 33863913
- [Derived] Smyth LM, Tamura K, Oliveira M, Ciruelos EM, Mayer IA, Sablin MP, Biganzoli L, Ambrose HJ, Ashton J, Barnicle A, Cashell DD, Corcoran C, de Bruin EC, Foxley A, Hauser J, Lindemann JPO, Maudsley R, McEwen R, Moschetta M, Pass M, Rowlands V, Schiavon G, Banerji U, Scaltriti M, Taylor BS, Chandarlapaty S, Baselga J, Hyman DM. Capivasertib, an AKT Kinase Inhibitor, as Monotherapy or in Combination with Fulvestrant in Patients with AKT1 E17K-Mutant, ER-Positive Metastatic Breast Cancer. Clin Cancer Res. 2020 Aug 1;26(15):3947-3957. doi: 10.1158/1078-0432.CCR-19-3953. Epub 2020 Apr 20. PMID 32312891
- [Derived] Banerji U, Dean EJ, Perez-Fidalgo JA, Batist G, Bedard PL, You B, Westin SN, Kabos P, Garrett MD, Tall M, Ambrose H, Barrett JC, Carr TH, Cheung SYA, Corcoran C, Cullberg M, Davies BR, de Bruin EC, Elvin P, Foxley A, Lawrence P, Lindemann JPO, Maudsley R, Pass M, Rowlands V, Rugman P, Schiavon G, Yates J, Schellens JHM. A Phase I Open-Label Study to Identify a Dosing Regimen of the Pan-AKT Inhibitor AZD5363 for Evaluation in Solid Tumors and in PIK3CA-Mutated Breast and Gynecologic Cancers. Clin Cancer Res. 2018 May 1;24(9):2050-2059. doi: 10.1158/1078-0432.CCR-17-2260. Epub 2017 Oct 24. PMID 29066505
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3610C00001&attachmentIdentifier=8eb42172-37bf-422c-a4b6-5f5da176091d&fileName=d3610c00001-revised-csp-10_redacted_SECURE.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3610C00001&attachmentIdentifier=82913ad8-331e-4f2e-9a50-9b31db606be3&fileName=d3610c00001_CSRSynopsis.pdf&versionIdentifier=